CLINICAL TRIAL: NCT02714855
Title: Apixaban in the Prevention of Stroke and Systemic Embolism in Patients With Atrial Fibrillation in Real-Life Setting in France - Cross-sectional Study
Brief Title: Apixaban in the Prevention of Stroke and Systemic Embolism in Patients With Atrial Fibrillation in Real-Life Setting in France
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-345
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Anticoagulation
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Apixaban

SUMMARY:
The present study will be conducted to assess the following research questions in real-life conditions in France:

What are the patient and disease characteristics, comorbidities and treatment history in NVAF patients initiating a new Anticoagulant (AC) treatment, according to treatment currently available and prescribed (apixaban, other NOACs, VKAs), and are the AC-naive patient profiles different from one treatment pattern to another when initiating a new AC treatment?

What are the HCP's reasons for discontinuing the previous AC strategy for initiating and choosing the newly initiated AC treatment in NVAF patients?

What are the conditions of newly-initiated apixaban prescriptions in NVAF patients: prescriber, proportion of naïve/experienced patients, daily dosage and number of daily doses?

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Diagnosed with non valvular atrial fibrillation (NVAF)
* Prescribed with a newly initiated AC treatment (apixaban, other NOACs or VKAs). Newly initiated AC treatment is defined as any AC treatment initiated within the past 3 months, including day of enrolment

Exclusion Criteria:

* Patients with atrial fibrillation (AF) due to reversible causes
* Patients with a diagnosis of VAF. The term VAF is used to imply that AF is related to rheumatic valvular disease (predominantly mitral stenosis) or prosthetic heart valves
* Patients participating in an ongoing clinical trial in AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiologists in france caring AF patients
Sampling Method: Probability Sample
Enrollment: 2081 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient characteristics in NVAF patients initiating a new AC-treatment | Approximately 12 months
  Patient's characteristics: age, gender, weight and height, BMI, dependence status
Comparing patient characteristics between apixaban and other Novel anticoagulants (NOACs) in AC-naive patients | Approximately 12 months
Comparing patient characteristics between apixaban and Vitamin K antagonists (VKAs) in AC-naive patients | Approximately 12 months
Disease characteristics in NVAF patients initiating a new AC-treatment | Approximately 12 months
  Disease characteristics: type of NVAF (permanent, paroxystic, persistent) ALD status (ALD: Affections de Longue Duree) for long term disease status (ALD 5, other ALDs specified, any ALD), disease duration
Comparing disease characteristics between apixaban and other NOACs in AC-naive patients | Approximately 12 months
Comparing disease characteristics between apixaban and VKAs in AC-naive patients | Approximately 12 months
Comorbidities in NVAF patients initiating a new AC-treatment | Approximately 12 months
  Comorbidities: congestive heart failure history, hypertension, diabetes mellitus, stroke/transient ischemic attack)/thromboembolism history, vascular disease history, renal impairment, liver impairment, prior major bleeding
Comparing comorbidities characteristics between apixaban and other NOACs in AC-naive patients | Approximately 12 months
Comparing comorbidities characteristics between apixaban and VKAs in AC-naive patients | Approximately 12 months
Treatment history in NVAF patients initiating a new AC-treatment | Approximately 12 months
  Treatment history: Previous AC strategy (no treatment, apixaban, other NOAC, VKAs) , Duration with previous AC strategy and indication of previous AC treatment
Comparing treatment history characteristics between apixaban and other NOACs in AC-naive patients | Approximately 12 months
Comparing treatment history characteristics between apixaban and VKAs in AC-naive patients | Approximately 12 months

SECONDARY OUTCOMES:
Distribution of previous AC strategy (no treatment, apixaban, other NOAC, VKAs) | Approximately 12 months
Distribution of reasons for discontinuing previous AC treatment among patients who had previous AC treatment | Approximately 12 months
  Reason(s) for discontinuing previous AC strategy (multiple choices accepted):
  Minor Bleeding event, major bleeding event, gastro-intestinal bleeding, dosing frequency, high bleeding risk, fear of side effect, cost and concern with renal function, dyspepsia, frequent falls or frailty, patient decision, concomitant treatment, concomitant chronic disease
Distribution of prescriber (Cardiologist him/herself, General Practitioner (GP), other) | Approximately 12 months
Distribution of reasons for initiating a new AC treatment | Approximately 12 months
Distribution of reasons for choosing the newly initiated AC treatment | Approximately 12 months
  Reason(s) for choosing the newly initiated AC treatment (multiple choices accepted):
  Physician preference, patient preference, results of a specific trial in relation to the clinical setting, cost and dosing frequency
Conditions of prescription of apixaban in NVAF patients | Approximately 12 months
  Condition of prescription of apixaban:
  Daily dosage (mg) at apixaban initiation, number of doses per day at apixaban initiation
Proportion of AC-naive patients | Approximately 12 months
Proportion of AC-experienced patients | Approximately 12 months
Mean daily dosage of daily doses for prescribed apixaban treatment according to patient characteristics | Approximately 12 months
Mean number of daily doses for prescribed apixaban treatment according to patient characteristics | Approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Fontaine-lès-Dijon, France

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx